CLINICAL TRIAL: NCT02682511
Title: A Phase 2 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Ifetroban in Patients With Diffuse Cutaneous Systemic Sclerosis (SSc) or SSc-associated Pulmonary Arterial Hypertension (SSc-PAH)
Brief Title: Oral Ifetroban to Treat Diffuse Cutaneous Systemic Sclerosis (SSc) or SSc-associated Pulmonary Arterial Hypertension
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-IFE-004
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Scleroderma, Diffuse; Scleroderma, Systemic; Scleroderma, Limited; Sclerosis, Progressive Systemic; Skin Diseases; Connective Tissue Diseases; Pathologic Processes; Autoimmune Diseases
Keywords: Ifetroban; Scleroderma; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Scleroderma, Limited; Skin Diseases; Connective Tissue Diseases; Pathologic Processes; Autoimmune Diseases | interventions — ifetroban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Patients with dcSSc (Experimental): Patients with dcSSc will be randomized to receive either oral ifetroban or oral placebo daily for 365 days
  Interventions: Drug: Oral Ifetroban; Drug: Oral Placebo
- Patients with SSc-PAH (Experimental): Patients with SSc-PAH will be randomized to receive either oral ifetroban or oral placebo daily for 365 days
  Interventions: Drug: Oral Ifetroban; Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Ifetroban — Subjects will be treated with oral ifetroban or placebo daily for 365 days
  Other Names: Ifetroban
Drug: Oral Placebo — Subjects will be treated with oral ifetroban or placebo daily for 365 days
  Other Names: Ifetroban

SUMMARY:
The purpose of this phase 2 multicenter, randomized, double-blind, placebo-controlled, study is to assess the safety and efficacy of ifetroban in patients with diffuse cutaneous systemic SSc (dcSSc) or SSc-associated pulmonary arterial hypertension (SSc-PAH).

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blind phase 2 trial of patients with dcSSc or SSc-PAH. Twenty participants with SSc-PAH and 14 participants with dcSSc will be randomized to receive either oral ifetroban daily or matching placebo. Study participants will be treated for 12 months, followed by a 30-day follow-up period. The study will test whether ifetroban is safe and statistically superior to placebo in reducing the effects of their disease at month 12 and explore the ability of ifetroban to prevent or reverse progression in patients with early disease duration and reverse established disease in patients with longer disease duration.

ELIGIBILITY:
Inclusion Criteria:

Diffuse Cutaneous Criterion:

1. Systematic Sclerosis (SSc), as defined using the 2013 American College of Rheumatology/ European Union League Against Rheumatism Classification Criteria and dcSSc within 7 years following initial diagnosis as defined by the onset of the first non-Raynaud symptom.

SSc-PAH Criteria:

1. Adults fulfilling the 2013 American College of Rheumatology/ European Union League Against Rheumatism Classification Criteria with confirmed SSc-PAH (limited or dcSSc) confirmed via previous cardiac catheterization
2. Stable oral therapy for PAH for at least 30 days (monotherapy or combination)
3. New York Heart Association (NYHA) Class I-III Heart Failure

Exclusion Criteria:

1. Have a diagnosis of systemic sclerosis sine scleroderma;
2. Be less than 18 years of age or greater than or equal to 80 years of age;
3. Be pregnant, nursing, or planning to become pregnant;
4. Current or planned treatment with prostanoid therapy;
5. Current or planned treatment with pirfenidone;
6. Use of rituximab in the last 3 months;
7. Use of mycophenolic acid (Myfortic, CellCept) at a stable dose for less than 3 months;
8. Current or planned corticosteroid therapy greater than 15mg per day of prednisone or prednisone equivalent;
9. Significant lung disease, defined as FVC < 50% predicted or DLCO <40% predicted;
10. Significant kidney disease, defined as Glomerular Filtration Rate (GFR) < 60 ml/min;
11. Have moderate or severe hepatic impairment;
12. Contraindication to MRI (e.g., implanted magnetic material, claustrophobia);
13. Known hypersensitivity to gadolinium;
14. Any cause of pulmonary hypertension other than World Health Organization (WHO) Group I associated with SSc;
15. Use of aspirin > 81 mg per day in the last two weeks;
16. Use of warfarin, heparin or other anticoagulants in the last 30 days;
17. Recent (within 6 weeks) myocardial infarction or persistent atrial arrhythmias;
18. Have a history of allergy or hypersensitivity to ifetroban;
19. Have taken investigational drugs within 30 days before study treatment administration;
20. Inability to understand the requirements of the study, inability to understand spoken English and abide by the study restrictions and to return for the required treatments and assessments;
21. Be otherwise unsuitable for the study, in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and Serious AEs (SAEs) | 56 weeks
  Safety is measured using AEs, including clinical significant changes in vital signs, laboratory test abnormalities and clinical tolerability of ifetroban.

SECONDARY OUTCOMES:
Change from baseline in forced vital capacity (FVC) | Baseline, 12, 26, and 52 weeks
  To determine if ifetroban improves pulmonary function in subjects with diffuse cutaneous SSc or SSc-PAH compared to placebo as measured by a change from baseline FVC.
Change from baseline in diffusion capacity for carbon monoxide (DLCO) | Baseline, 12, 26, and 52 weeks
  To determine if ifetroban improves pulmonary function in subjects with diffuse cutaneous SSc or SSc-PAH compared to placebo as measured by a change from baseline diffusion capacity for carbon monoxide (DLCO)
Change from baseline in the modified Rodnan skin score (mRSS) | Baseline, 12, 26, 39, and 52 weeks
  The efficacy of treatment on skin fibrosis will be measured by changes from baseline in mRSS, a measure of skin thickness, at 52 weeks.

OTHER OUTCOMES:
Change from baseline in ventricular function as determined by cardiac MRI | Baseline, 26, and 52 weeks
Change from baseline in ventricular function as determined by echocardiography | Baseline, 26, and 52 weeks
Improve skin and peripheral vascular disease as measured by active digital ulcer count | Baseline, 12, 26, 39, and 52 weeks
Improve skin and peripheral vascular disease as measured by the subject's self-assessment of pain in digits by a visual analog scale (VAS), if active digital ulcers are present. | Baseline, 12, 26, 39, and 52 weeks
Change from baseline in blood biomarkers | Baseline, 26, and 52 weeks
Change from baseline in skin biomarkers | Baseline, 26, and 52 weeks
Change from baseline in erythrocyte sedimentation rate | Baseline, 26, and 52 weeks
Change from baseline in subject-reported health status assessed by the Scleroderma Health Assessment Questionnaire (SHAQ) | Baseline, 12, 26, 39, and 52 weeks
Change from baseline in subject health and disability measurements as assessed by the World Health Organization Disability Assessment Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, 12, 26, 39, and 52 weeks
Change from baseline in subject-reported gastro-intestinal tract symptoms as assessed by the University of California, Los Angles (UCLA) Scleroderma Clinical Trial Consortium (SCTC) Gastrointestinal Tract (GIT) Questionnaire | Baseline, 12, 26, 39, and 52 weeks
Change from baseline in subject-reported outcomes as assessed by the short-form health survey (SF-36) | Baseline, 12, 26, 39, and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Evan Brittain, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (13):
- United States (10):
  - The Universtity of Arizona Arthrtis Center, Tucson, Arizona
  - UCLA, Los Angeles, California
  - Cleveland Clinic - Florida, Weston, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Research Institute, Dallas, Texas
- India (3):
  - PGIMER, Chandigarh, Chandigarh
  - KDH - Kokilaben Dhirubhai Ambani Hospital, Mumbai, Maharashtra
  - B. J. Government Medical College, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No